CLINICAL TRIAL: NCT02009215
Title: 'SCHOOL-BASED TREATMENT WITH ACT TO REDUCE TRANSMISSION' (START-IPT): Evaluation of the Community Impact of Intermittent Preventive Treatment for Malaria in Ugandan Children: a Cluster Randomised Trial
Brief Title: School-Based Treatment With ACT to Reduce Transmission
Acronym: START-IPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Infectious Diseases Research Collaboration, Uganda (Other); University of California, San Francisco (Other); University of Durham (Other)
Responsible Party: Principal Investigator, Sarah Staedke, Principal Investigator, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ITCRAA6910
Record Dates: First submitted 2013-10-23; First posted 2013-12-11 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Malaria
Keywords: Uganda; intermittent preventive treatment; dihydroartemisinin-piperaquine; schoolchildren; malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intermittent preventive treatment (IPT) (Experimental): Dihydroartemisinin-piperaquine (DP)
  Interventions: Drug: Dihydroartemisinin-piperaquine (DP)
- Control (No Intervention): No intermittent preventive treatment (IPT) with dihyroartemisinin-piperaquine (DP) will be given.

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine (DP) — Intermittent preventive treatment (IPT) with dihyroartemisinin-piperaquine (DP) will be delivered to participating students monthly, for up to 6 rounds of treatment during one school year. DP will be given once a day for 3 days, using full strength tablets (40/320mg) according to weight-based guidelines. Treatment will be directly observed, and will not be blinded.
  Other Names: Duo-cotecxin
  Arms: Intermittent preventive treatment (IPT)

SUMMARY:
We propose to evaluate the community-level impact of intermittent preventive treatment (IPT) for malaria in schoolchildren on clinical outcomes and malaria transmission, using a cluster-randomised design in Jinja, Uganda. Dihydroartemisinin-piperaquine (DP) will be administered to schoolchildren monthly for up to six rounds of treatment during one school year. Outcomes will be measured using surveys of communities, schoolchildren, and mosquito vectors. Our proposal also includes health service research to evaluate the potential feasibility of taking the programme to scale, which will guide future research and implementation of the intervention, and help shape policies in Uganda and elsewhere in Africa.

DETAILED DESCRIPTION:
Study objective: The primary objective of the study is to evaluate the impact of IPT for malaria in schoolchildren using monthly DP, as compared with the current standard of care (no IPT), on community-level indicators of malaria transmission. We will test the hypothesis that malaria transmission, as measured by the prevalence of asexual parasitaemia and the entomological inoculation rate (EIR), will be lower in communities surrounding the intervention schools, than those surrounding the control schools.

Study site: The study will be conducted in Jinja district, Uganda.

Clusters: A cluster will be defined as one primary day school plus the 100 closest households surrounding the school. The clusters will be defined prior to randomisation using digitally enumerated maps. We plan to include approximately 84 clusters in the study, with one school per cluster; half will be randomised to the IPT intervention, and half to control.

Randomisation: Randomisation will be conducted by the trial statistician, who is not directly involved in the field activities. Primary schools will be stratified by type of ownership (public vs private). Restricted randomisation will be employed to ensure balance on type of school and geographical location.

Study population: The intervention will be delivered to children attending participating primary schools that are randomised to the intervention group.

The IPT intervention: IPT with dihydroartemisinin-piperaquine (DP) will be delivered to all schools located in the intervention clusters. Treatment will be administered to participating students monthly, for up to 6 rounds of IPT during one school year, and will not be blinded.

Administration of DP: All enrolled students will receive DP (Duo-cotexcin, Holley Cotec Pharmaceuticals) given once a day for 3 consecutive days. DP will be dosed according to weight-based guidelines. Full-strength DP tablets (40/320mg) will be administered orally by study personnel, and all treatments will be directly observed.

Evaluation procedures: Outcomes will be measured through surveys of communities, schoolchildren, and mosquito vectors. In addition, the safety of IPT with monthly DP, and the potential feasibility of the IPT intervention will also be assessed.

1. Community surveys. Cross-sectional surveys of community residents living in households randomly selected from each cluster will be conducted at baseline and at the end of intervention.The community surveys will consist of two components: (1) a household survey questionnaire administered to heads of households, and (2) a clinical survey including laboratory testing of all household residents. The primary outcome of the community surveys will be parasite prevalence as measured by microscopy. In the final community survey, we plan to enroll 105 participants per cluster (8820 total).
2. School surveys. Cross-sectional surveys of students randomly selected from each cluster school will be conducted at baseline and at the end of intervention. The primary outcome of the school surveys will be parasite prevalence as measured by microscopy. In the final school survey, we plan to enroll 13 students per cluster (1092 total).
3. Entomology surveys. Mosquitos will be collected using Centers of Disease Control and Prevention (CDC) light traps from 5 randomly selected households from 20 clusters in each study arm (100 households per arm, 200 total), using a list randomly generated from the enumeration database. Each house will be sampled once a month for the duration of the study. The primary outcome of the entomology surveys will be EIR.
4. Safety monitoring. Students enrolled in the intervention will be evaluated prospectively for serious adverse events. To assess the impact of monthly IPT with DP on risk of cardiotoxicity, a sub-set of participants (n=189) will be selected using convenience sampling (from the intervention arm only) to participate in cardiac monitoring and a pharmacokinetic study.
5. Qualitative assessment. A qualitative study will run alongside the main trial, to investigate the potential feasibility for integrating this intervention into routine health services and school systems. We will conduct a historical review of published and unpublished literature on programmes that have integrated health interventions into the education sector; ethnographic observation of intervention activities; and in-depth interviews with key stakeholders, and teachers and health workers.

Analytical plan

1. Quantitative surveys: All data will be analysed on the basis of intention-to-treat, that is, community residents and school children taking part in the final surveys will be classified as participating in the intervention or control according to the randomization assignment of the cluster they were surveyed in, regardless of whether they (or their children) received the intervention or not. The primary outcome is prevalence of asexual parasitaemia in the community surveys. Prevalence of asexual parasitaemia in the school surveys and EIR are secondary outcome measures. An individual-level approach to the analysis will be used due to the large number of clusters per arm.

   For binary outcomes, generalised linear Poisson models with log link function will be used. The effect of the intervention will be quantified by calculation of a prevalence risk ratio. For quantitative outcomes, linear regression models will be used. The effect of the intervention will be quantified by calculation of difference in mean outcome. Rate ratios will be used to describe the effect of the intervention on rates. An estimate of the coefficient of variation, k, will be provided overall and for the community survey for each age group (as defined by the stratified sampling).

   The probability of selection for the final community survey was related to the sampling frame which was determined by the expected parasite prevalence (which varies by age) in age categories; < 5 years, 5-15 years, > 15 years. Therefore, the age structure of the study population is not representative of the community population as a whole. Because we are looking at the community effect we will use inverse probability weights based on the age population structure of all clusters as recorded by the census survey. In practice, each individual will be assigned one of three weights, generated using the census survey, and based on their age as recorded at the final community survey. Population estimates of prevalence will be obtained using svy commands with the cluster as the primary sampling unit and age-related inverse probability weights. Children selected for the school survey were randomly selected after stratification by class. Households selected for the entomological survey were also randomly selected. No weighting is therefore required for the analysis of either the school or entomological surveys.

   The effect of the intervention will also be assessed using adjusted analyses. The cluster-specific prevalence or mean from the baseline survey will be adjusted for where available. Variables collected in the baseline community survey, which were imbalanced between trial arms, and likely to be prognostic for outcomes will be adjusted for. Secondary analyses will be conducted to assess whether the effect of the intervention differs by age group or school type. The effect of the intervention for each outcome will be examined by age group or school type and tests for interaction conducted.
2. Qualitative data: The data analysis of the field notes and in-depth interviews will follow a bottom-up approach, identifying repeating patterns in the data. Field notes will be coded on a daily basis using qualitative data analysis software, NVivo (QSR International, Cambridge, MA). Transcripts will be coded line-by-line, and then later developing themes and theoretical constructs by grouping the base coding together. A coding template will be developed and refined. Following the coding process, themes and theoretical constructs will be developed from both the field notes and the interview transcripts, and the analysis will be conducted with reference to the literature and theory regarding school-based and cross-sectoral interventions. Following this analysis, the interpretation will take on an applied stance, to seek out specific challenges and opportunities for methods and content of interventions to support implementation of IPT.

ELIGIBILITY:
For IPT intervention

Inclusion Criteria:

1. Student enrolled in a participating intervention school.
2. Willingness of parent/guardian to provide written informed consent.
3. Provision of written assent by the student (aged 8 years or above).

Exclusion Criteria:

1. Age < 5 years
2. Known allergy or history of adverse reaction to DP
3. Menarche in female students
4. Weight < 11 kg
5. History of cardiac problems or fainting
6. Family history of long QT syndrome
7. Current use of medications known to prolong the QT interval
8. Not able to locate parent or guardian, after at least three attempts including parent/teacher association (PTA) meetings and home visits
9. Not able to locate the student at school, after at least three attempts

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10746 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Parasite prevalence measured by microscopy in final community survey | Approximately 1-4 months after completion of the intervention
  Proportion of thick blood smears that are positive for asexual parasites, as measured by microscopy.

SECONDARY OUTCOMES:
Entomologic inoculation rate (EIR) in the entomology survey | Over approximately 1 year
  EIR will be defined as the number of infectious bites per person per year (the human biting rate multiplied by the sporozoite rate).
Parasite prevalence measured by microscopy in the final school survey | During the final 1 month of the intervention
  Proportion of thick blood smears that are positive for asexual parasites, as measured by microscopy.

OTHER OUTCOMES:
Parasite prevalence measured by microscopy + LAMP in the final community survey | Approximately 1-4 months after completion of the intervention
  Proportion of samples that are positive for asexual parasites by microscopy and LAMP
Prevalence of anaemia in children under-five in the final community survey | Approximately 1-4 months after completion of the intervention
  Proportion of haemoglobin measurements categorised as mild, moderate, and severe anaemia according to WHO age-stratified guidelines, in children under five
Prevalence of gametocytaemia in the final community survey | Approximately 1-4 months after completion of the intervention
  Proportion of thick blood smears that are positive for sexual parasites
Sporozoite rate in the entomology survey | Over approximately 1 year
  Proportion of An gambiae infected with sporozoites
Prevalence of serious adverse events (SAEs) | Over approximately 6 months, during the delivery of the intervention
  Proportion of children enrolled in the intervention experiencing any SAEs out of the total number of children enrolled; collected during prospective monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Sarah G Staedke, MD, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Infectious Diseases Research Collaboration, Kampala, Uganda

REFERENCES:
- [Background] Nankabirwa J, Cundill B, Clarke S, Kabatereine N, Rosenthal PJ, Dorsey G, Brooker S, Staedke SG. Efficacy, safety, and tolerability of three regimens for prevention of malaria: a randomized, placebo-controlled trial in Ugandan schoolchildren. PLoS One. 2010 Oct 19;5(10):e13438. doi: 10.1371/journal.pone.0013438. PMID 20976051
- [Background] Nankabirwa JI, Wandera B, Amuge P, Kiwanuka N, Dorsey G, Rosenthal PJ, Brooker SJ, Staedke SG, Kamya MR. Impact of intermittent preventive treatment with dihydroartemisinin-piperaquine on malaria in Ugandan schoolchildren: a randomized, placebo-controlled trial. Clin Infect Dis. 2014 May;58(10):1404-12. doi: 10.1093/cid/ciu150. Epub 2014 Mar 12. PMID 24621953
- [Derived] Rehman AM, Maiteki-Sebuguzi C, Gonahasa S, Okiring J, Kigozi SP, Chandler CIR, Drakeley C, Dorsey G, Kamya MR, Staedke SG. Intermittent preventive treatment of malaria delivered to primary schoolchildren provided effective individual protection in Jinja, Uganda: secondary outcomes of a cluster-randomized trial (START-IPT). Malar J. 2019 Sep 18;18(1):318. doi: 10.1186/s12936-019-2954-0. PMID 31533845
- [Derived] Staedke SG, Maiteki-Sebuguzi C, Rehman AM, Kigozi SP, Gonahasa S, Okiring J, Lindsay SW, Kamya MR, Chandler CIR, Dorsey G, Drakeley C. Assessment of community-level effects of intermittent preventive treatment for malaria in schoolchildren in Jinja, Uganda (START-IPT trial): a cluster-randomised trial. Lancet Glob Health. 2018 Jun;6(6):e668-e679. doi: 10.1016/S2214-109X(18)30126-8. Epub 2018 Apr 13. PMID 29661635
- See also: Infectious Disease Research Collaboration (IDRC), Uganda Malaria Surveillance Project (UMSP), Makerere University - University of California, San Francisco (MU-UCSF) — http://www.muucsf.org